CLINICAL TRIAL: NCT03164304
Title: Efficacy and Safety of One Gram Versus Two Grams Intravenous Maintenance Dose of Magnesium Sulfate in Women With Severe Pre-eclampsia: a Randomized Clinical Trial.
Brief Title: Efficacy and Safety of 1 g Vs 2 g Per Hour Intravenous Maintenance Dose of MgSO4 in Women With Severe Pre-eclampsia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1g vs 2g MgSO4
Record Dates: First submitted 2017-05-17; First posted 2017-05-23 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Severe Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Magnesium Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One gram magnesium sulfate (Active Comparator): Pregnant women with a diagnosis of severe pre-eclampsia will receive 1 g of mgso4 to prevent and control of convulsions
  Interventions: Drug: Magnesium Sulfate
- Two grams magnesium sulfate (Experimental): Pregnant women with a diagnosis of severe pre-eclampsia will receive 2 g of mgso4 to prevent and control of convulsions
  Interventions: Drug: Magnesium Sulfate

INTERVENTIONS:
Drug: Magnesium Sulfate — intravenous

SUMMARY:
Preeclampsia is commonly viewed as one of the hypertensive pregnancy disorders, which cover a spectrum of clinical presentations from chronic hypertension ( hypertension occurring prior to 20 weeks of gestation) and gestational hypertension (hypertension occurring after 20 weeks of gestation) To more severe forms, including preeclampsia, eclampsia (its convulsive form), and HELLP syndrome (hemolysis, elevated liver enzyme S, and low platelets)

DETAILED DESCRIPTION:
Treatment for patients who have developed preeclampsia or eclampsia mainly consists of control of hypertension, magnesium sulphate for prevention of eclampsia and convulsions, and planning for delivery.

Magnesium sulfate has been used to prevent eclamptic convulsion since 1925, its efficacy was confirmed by a large randomized controlled trial in 2002. Eclampsia could be prevented in more than 50% after magnesium sulfate administration . The World Health Organization recommended magnesium sulfate as the most effective, safe, and low-cost drug for the prevention of seizure in severe preeclampsia and eclampsia . The recommended dose of magnesium sulfate is 4 to 6 gram intravenous loading dose, followed by maintenance intravenous drip at the rate of 1 to 2 gram per hour .

Although different magnesium sulfate regimens have been tested, two dosing regimens are internationally recommended and widely used. The Pritchard regimen is a predominantly intramuscular regimen given as a loading dose of 4 g intravenously , and 5 g Intramuscular into each buttock followed by a maintenance dose of 5 g Intramuscular every 4 hours. This regimen is popular in resource-limited settings where intravenously administration of magnesium sulfate may not be feasible. However, it is associated with pain and a higher risk of infection at the injection site.

The Zuspan regimen is given as a 4 gram intravenously loading dose followed by continuous intravenously infusion of 1 gram per hour.

Either 1 gram or 2 gram maintenance dose of Magnesium Sulphate has been reported to reduce the development of eclampsia. Randomized controlled trials offering direct comparison between these 2 doses are lacking.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women admitted to Women health hospital with a diagnosis of severe pre-eclampsia

Exclusion Criteria:

* 1- Women with Non-proteinuric hypertension, 2- severe renal impairment 3- Myasthenia gravis 4- High amount of magnesium in blood 5- Low or high amount of calcium in blood 6- Myocardial damage, diabetic coma, heart block

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
The rate of convulsions in each group. | 24 hour
  the number of participants who have convulsion
The percentage of women reaching the Mg therapeutic level of 4,8 mg/dl | 24 hour
  Follow up by Serum Magnesium level
The rate of adverse events in each group | 24 hour
  the number of participants who have adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, woman health hospital, Asyut, Egypt

REFERENCES:
- [Background] Altman D, Carroli G, Duley L, Farrell B, Moodley J, Neilson J, Smith D; Magpie Trial Collaboration Group. Do women with pre-eclampsia, and their babies, benefit from magnesium sulphate? The Magpie Trial: a randomised placebo-controlled trial. Lancet. 2002 Jun 1;359(9321):1877-90. doi: 10.1016/s0140-6736(02)08778-0. PMID 12057549
- [Background] Zakiyah N, Postma MJ, Baker PN, van Asselt AD; IMPROvED Consortium. Pre-eclampsia Diagnosis and Treatment Options: A Review of Published Economic Assessments. Pharmacoeconomics. 2015 Oct;33(10):1069-82. doi: 10.1007/s40273-015-0291-x. PMID 26048352
- [Background] Hypertension in pregnancy. Report of the American College of Obstetricians and Gynecologists' Task Force on Hypertension in Pregnancy. Obstet Gynecol. 2013 Nov;122(5):1122-1131. doi: 10.1097/01.AOG.0000437382.03963.88. No abstract available. PMID 24150027
- [Derived] Diaz V, Long Q, Oladapo OT. Alternative magnesium sulphate regimens for women with pre-eclampsia and eclampsia. Cochrane Database Syst Rev. 2023 Oct 10;10(10):CD007388. doi: 10.1002/14651858.CD007388.pub3. PMID 37815037